CLINICAL TRIAL: NCT05417958
Title: A Novel N-of-1 Randomized, Controlled, Clinical Trial to Assess the Effect of Blenderized Tube Feeds on Esophagogastric Physiology
Brief Title: Clinical Trial of Blenderized Tube Feeds Varying in Viscosity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Bridget Hron, Staff Physician, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00042262
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Feeding Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Extremely Thick - Mildly Thick - Extremely Thick - Mildly Thick (Experimental): Participants will receive 4 weeks Extremely Thick, 4 weeks Mildly Thick, 4 weeks Extremely Thick and 4 weeks Mildly Thick blenderized tube feeds. The volume, caloric density and frequency will be matched to pre-study feeding regimen.
  Interventions: Other: Extremely thick blenderized tube feed; Other: Mildly thick blenderized tube feed
- Extremely Thick - Mildly Thick - Mildly Thick - Extremely Thick (Experimental): Participants will receive 4 weeks Extremely Thick, 4 weeks Mildly Thick, 4 weeks Mildly Thick and 4 weeks Extremely Thick blenderized tube feeds. The volume, caloric density and frequency will be matched to pre-study feeding regimen.
  Interventions: Other: Extremely thick blenderized tube feed; Other: Mildly thick blenderized tube feed
- Mildly Thick - Extremely Thick - Extremely Thick - Mildly Thick (Experimental): Participants will receive 4 weeks Mildly Thick, 4 weeks Extremely Thick, 4 weeks Extremely Thick and 4 weeks Mildly Thick blenderized tube feeds. The volume, caloric density and frequency will be matched to pre-study feeding regimen.
  Interventions: Other: Extremely thick blenderized tube feed; Other: Mildly thick blenderized tube feed
- Mildly Thick - Extremely Thick - Mildly Thick - Extremely Thick (Experimental): Participants will receive 4 weeks Mildly Thick, 4 weeks Extremely Thick, 4 weeks Mildly Thick and 4 weeks Extremely Thick blenderized tube feeds. The volume, caloric density and frequency will be matched to pre-study feeding regimen.
  Interventions: Other: Extremely thick blenderized tube feed; Other: Mildly thick blenderized tube feed

INTERVENTIONS:
Other: Extremely thick blenderized tube feed — Commercial blenderized tube feed, not diluted
Other: Mildly thick blenderized tube feed — Commercial blenderized tube feed, diluted with ingredients contained in blend

SUMMARY:
The investigators are conducting a 16 week multiple cross-over study (N-of-1 trial) comparing two blenderized tube feeds varying in viscosity in 40 children.

ELIGIBILITY:
Inclusion Criteria:

* age > 1 year
* >90% of total calories via G-tube for > 6 months
* G-tube diameter ≥ 14 French
* moderate severity of upper GI symptoms of nausea, bloating, postprandial fullness and early satiety defined as Gastroparesis Cardinal Symptom Index-Daily Diary (GCSI-DD) composite score > 2
* anticipated stable GI-related medications for the duration of the study.

Exclusion Criteria:

* cystic fibrosis, primary ciliary dyskinesia, interstitial lung disease, bronchiolitis obliterans, or lung transplant
* untreated malabsorptive intestinal disease (e.g. Crohn's disease, celiac disease)
* Nissen fundoplication
* use of non-standard enteral formulas (e.g. ketogenic formulas) for the management of metabolic, endocrine or neurologic rare diseases
* allergy or intolerance to any component of the study diet
* inability to tolerate bolus gastric feeds.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Upper GI symptoms | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  differences in daily parental rating of upper gastrointestinal symptoms from the validated Gastroparesis Cardinal Symptom Index-Daily Diary (GCSI-DD) between extremely and mildly thick blenderized tube feeds

SECONDARY OUTCOMES:
Gastrointestinal symptoms | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptoms Questionnaire, scale of 0 to 100, higher scores indicate less symptom burden
Gastrointestinal symptoms | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  Pediatric Quality of Life Inventory Gastroparesis Questionnaire, , scale of 0 to 100, higher scores indicate less symptom burden
Pulmonary symptoms | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  Pediatric Cough Questionnaire, score ranges from 0 to 25, higher scores indicate less symptom burden
Health care utilization | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  frequency of hospital admissions
Health care utilization | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  length of hospital admissions
Health care utilization | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  rates of ER/urgent care visits
GI medication use | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  % of participants requiring acid suppressive medication or GI motility agents such as cyproheptadine and erythromycin
Height | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  height
Weight | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  Weight or weight for length
Weight for height/body mass index (BMI) | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  weight for height (children < 2) or BMI (over 2 years of age)
number of patients with unplanned G-tube exchange | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
urine output adequacy | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  frequency of urine output
rate of respiratory suctioning per day | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  how often suctioning is required (e.g. number of times per day)
need for antibiotics for pneumonitis | 8 weeks of extremely vs. 8 weeks of mildly thick blends (multiple cross-over design)
  frequency of antibiotics prescribed for pulmonary indications

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No